CLINICAL TRIAL: NCT06399536
Title: Individualized Acute Normovolemic Hemodilution for Non-cardiac Surgery With Anticipated High-dose Red Cells Transfusion
Brief Title: Individualized ANH for Non-cardiac Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Ren Liao, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WCH20240429
Record Dates: First submitted 2024-04-29; First posted 2024-05-03 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Transfusion Related Complication; Hemodilution
Keywords: acute normovolemic hemodilution; individualized blood transfusion; clinical trial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The clinical investigators, the responsible anesthesiologists and surgeons, the research assistants, and the participants will not be blinded to the treatment assignment, and the statisticians responsible for outcome analysis will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ANH group (Experimental): Participants will undergo individualized ANH based on the West China Liu's Score after anesthetic induction. The decision of autologous blood transfusion or allogeneic red cell transfusion will be made according to the West China Liu's Score.
  Interventions: Procedure: Individualized ANH
- Control group (No Intervention): Participants will be treated as the routine clinical practice. The decision of blood transfusion will be guided as the transfusion guideline.

INTERVENTIONS:
Procedure: Individualized ANH — Participants will undergo individualized ANH based on the West China Liu's Score after anesthetic induction. The decision of autologous blood transfusion or allogeneic red cell transfusion will be made according to the West China Liu's Score.
  Arms: ANH group

SUMMARY:
In this trial, we proposed an individualized acute normovolemic hemodilution (ANH), and conduct a randomized controlled trial to testify the effect of individualized ANH on red cells requirement for non-cardiac surgeries with anticipating major blood loss in adults.

DETAILED DESCRIPTION:
Allogeneic blood transfusion (ABT) is often given for patients undergoing major surgery with large amount of blood loss. However, ABT itself is associated with various complications, such as anaphylaxis, transfusion related bacterial and viral infections, and transfusion related lung injury [1-3]. Strategies for reduction of requirements for ABT during surgery continue to be of an importance in clinical practice.

The current strategies for ABT reduction during major surgery can be divided into the decrease of operative blood loss and the provision of autologous red cells. Collection of autologous red cells could be performed several weeks before admission (preoperative autologous donation, PAD), after anesthetic induction and prior to the surgical incision (acute normovolemic hemodilution, ANH), or during the operation (cell saver) [4]. ANH is a technique that remove the whole blood and infuse the colloids or crystalloids at the same time to get the hemodilution with the normal volume [5]. With the hemodilution, the amounts of red cells lost with bleeding could be reduced during surgery, and blood viscosity could be decreased beneficial for improved blood flow and increased venous return at a relative constant atrial pressure [6]. However, ANH has not been a widely accepted technique despite these advantages. One possible reason could be the mixed results about application of ANH in the literature. It was reported to decrease the risk of ABT when compared with the control group in a meta-analysis including 29 randomized controlled trials [7], but other authors reported ANH could only decrease intraoperative ABT with no differences in overall perioperative transfusion requirements [8]. Another reason could be due to the staffing shortage in clinical practice, especially in China. The implementation of AHN in the operating room requires the cooperation of a staff team including anesthesiologists, circulating nurses, and technicians from department of blood transfusion to collect the autologous blood and store it in refrigerators, and reinfuse the autologous blood under the supervision and double verification. In addition, what degree of the hemodilution should be achieved for a patient is lack of evidence and guidance, and the hemodilution can't be individualized executed.

In our previous study, we proposed the West-China-Liu's Score (Table.1) for individualized transfusion of red cells and conducted a multi-centered RCT to verify that the application of this individualized transfusion strategy can decrease the requirement of perioperative red cells transfusion when compared with the restrictive or liberal strategies without increase of complications in elective noncardiac surgeries [9]. According to the score, we can determine the tolerable lower level of hemoglobin (Hb), and it's safe for a patient to keep his Hb level above the score. With the West-China-Liu's Score, we dilute the patient's Hb level to the degree of the score plus 2, we can calculate the volume of the collected autologous blood. For example, a patient's initial Hb level is 12g/dL, the West-China-Liu's Score is 6, we dilute the Hb level to the score of 6+2=8, and the hemodilution level for him is Hb of 8g/dL. A 1g/dL Hb level is about 400ml of blood, and the decrease of Hb level from 12g/dL to 8g/dL is about 1600ml of blood. While we infuse the patient with fluids and collect blood at the same time, we will collect 800ml of the autologous blood for this patient. The collected autologous blood will be transfused to the patient when his Hb level is decreased to 6g/dL, or at the end of the operation. By this mean, ANH could be individualized.

Based on previous findings and the theory of individualized transfusion strategy, we hypothesize that individualized ANH under guidance of West-China Liu's Score can reduce the requirement of allogeneic red cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective non-cardiac surgery with an anticipated red blood cells transfusion >8 units (or 1600ml)
* Aged 18~75 years
* Preoperative Hb level > 120g/L for men and > 110g/L for women.

Exclusion Criteria:

* Refusal of blood transfusion
* Cardiopulmonary insufficiency
* Cerebrovascular disease
* Renal impairment
* Hemoglobinopathies or blood system diseases
* Other situations not suitable for inclusion in clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
ABT requirement | Up to 12 weeks.
  The perioperative allogeneic red blood cells consumption (Units per person).

SECONDARY OUTCOMES:
Proportion of transfused participants | Up to 12 weeks.
  The proportion of participants receiving allogeneic red blood cells.
Composite of in-hospital complications | Up to 12 weeks.
  The complications will be divided into five grades. Grade Ⅰ, recovery after temporary treatment, e.g., postoperative nausea and vomiting. Grade Ⅱ, prolonged hospitalization, e.g., infection requiring antibiotics treatment. Grade Ⅲ, life threatening complications requiring intense treatment during hospitalization, e.g., postoperative bleeding requiring re-operation, or acute renal insufficiency requiring dialysis therapy. Grade Ⅳ, life threatening complications resulting in significantly decreased quality of life, e.g., myocardial infarction. Grade Ⅴ, all-cause mortality during hospitalization.
Length of hospital stay | Up to 12 weeks.
  The time from the day of admission to discharge from the hospital (Unit: days).
Postoperative hospital stay | Up to 12 weeks.
  The time from the day of surgery to discharge from the hospital (Unit: days).
Total in-hospital cost | Up to 12 weeks.
  Total in-hospital cost

CONTACTS AND LOCATIONS:
Overall Officials: Ren Liao, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) with anonymity will be uploaded to the IPD sharing platform for data sharing. Data will be available after the agreement of the correspondence author upon reasonable request.
Supporting Information: Study Protocol, CSR
Time Frame: 5 years after the completion of the study.
Access Criteria: Upon request by email to PI.

REFERENCES:
- [Derived] Liao C, Tan J, An J, Zhong J, Lai X, Tian L, Liao R. Individualised acute normovolaemic haemodilution for non-cardiac surgery with anticipated high-dose red cell transfusion: study protocol for a randomised controlled trial in West China Hospital of Sichuan University. BMJ Open. 2025 Jan 2;15(1):e088326. doi: 10.1136/bmjopen-2024-088326. PMID 39753262